CLINICAL TRIAL: NCT02601768
Title: Occluder Size Determination in Transcatheter Closure of Ostium Secundum Atrial Septal Defect Based on Three-Dimensional Echocardiography Assessment
Brief Title: Occluder Size Determination in Transcatheter ASD II Closure Based on 3D TEE Assessment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: 2.11/VI/15
Record Dates: First submitted 2015-11-09; First posted 2015-11-10 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Ostium Secundum Atrial Septal Defect
Keywords: ASD II; transcatheter closure; percutaneous closure; 3D TEE; balloon-sizing
MeSH Terms: conditions — Heart Septal Defects, Atrial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ASD II: Transcatheter closure of ASD II
  Interventions: Device: Transcatheter closure of ASD II

INTERVENTIONS:
Device: Transcatheter closure of ASD II — Transcatheter closure of ASD II performed in our center.

SUMMARY:
The aim of this study is to determine whether three-dimensional tranesophageal echocardiography (3D TEE) assessment of ostium secundum atrial septal defect (ASD II) may be as efficient as two-dimensional (2D) TEE assessment complemented by the balloon-sizing during transcatheter closure of the defect.

DETAILED DESCRIPTION:
A total of 50 consecutive patients eligible to percutaneous ASD II closure will be enrolled in the study. 3D-TEE will be performed in the diagnostic process; the images will be recorded for further investigation, however, measurments of the defect will not be taken until after the procedure. Traditional 2D-TEE together with balloon-sizing assessment of the defect will be performed in enrolled patients in order to chose a device. Control transthoracic echocardiography (TTE) will be provided twice to evaluate the outcome of transcatheter treatment: 1 day after the procedure and 6-12 months later. The previously obtained 3D images will be retrospectively assessed by 2 independent investigators excluded from the interventionalists' team. Maximum and minimum diameter, perimeter and area of the defect will be measured to propose the assumed optimal occluder size. Correlation between proposed occluder size and the device used during the procedure will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* ASD II suitable for percutaneous treatment
* free and informed consent to analyze the medical data of the person concerned
* age: patients over 16

Exclusion Criteria:

* ASD II not suitable for percutaneous treatment
* any valvular heart disease requiring cardiac surgery
* no free and informed consent to analyze the medical data of the person concerned
* age: under 16

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 50 consecutive adult patients with ASD II closed percutaneously in our center in the study time frame i.e.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between the proposed and actual device size. | 18 months
  The correlation will be analyzed after the data of the whole group has been completed.

SECONDARY OUTCOMES:
Success rate of the procedure | 12 months
  Localization of the occluder in two echocardiographic assessments, 1 day and 6-12 months after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Henzel, MD, Study Director — Institute Of Cardiology in Warsaw
Locations (1):
- Institute Of Cardiology, Warsaw, Poland